CLINICAL TRIAL: NCT01672775
Title: A Phase 1, Open Label, Multi-center Study to Assess the Safety, Pharmacokinetics and Effectiveness of AGS-16C3F Monotherapy in Subjects With Renal Cell Carcinoma (RCC) of Clear Cell or Papillary Histology
Brief Title: A Study to Assess the Safety, Pharmacokinetics and Effectiveness of AGS-16C3F Monotherapy in Subjects With Renal Cell Carcinoma (RCC) of Clear Cell or Papillary Histology
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-16C3F-12-2
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Renal Cell; Renal Cell Carcinoma of Papillary Histology; Renal Cell Carcinoma With Clear Cell Histology; Renal Cell Carcinoma With Non-Clear Cell Histology
Keywords: Renal Cell Carcinoma; AGS-16C3F; Pharmacokinetics of AGS-16C3F
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — AGS-16C3F

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 AGS-16C3F highest dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- Cohort 0 AGS-16C3F higher dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- Cohort (-1) AGS-16C3F high dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- Cohort (-2) AGS-16C3F middle dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- Cohort (-3) AGS-16C3F low dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- Cohort (-4) AGS-16C3F lowest dose (Experimental): Renal Cell Carcinoma subjects with clear and non-clear histology
  Interventions: Drug: AGS-16C3F
- AGS-16C3F in RCC Subjects with Clear Cell Histology (Experimental): Expansion Cohort
  Interventions: Drug: AGS-16C3F
- AGS-16C3F in RCC Subjects with Papillary Histology (Experimental): Expansion Cohort
  Interventions: Drug: AGS-16C3F

INTERVENTIONS:
Drug: AGS-16C3F — intravenous (IV) infusion

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics and assess the immunogenicity and effectiveness of AGS-16C3F in subjects with renal cell cancer (RCC).

DETAILED DESCRIPTION:
The study has two components. The first aims to establish a safe dose for AGS-16C3F. Once identified, the safety and effectiveness will be tested in additional subjects with either clear cell or papillary histology in expanded cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Dose determination cohorts: Histologically confirmed diagnosis of metastatic RCC of either clear cell or non-clear histology.

  * Tumors with clear cell histology: subject must have progressed after at least one anti-vascular endothelial growth factor receptor (anti-VEGFR) therapy
  * Tumors with non-clear cell histology must be ectonucleotide pyrophosphatase/phosphodiesterase family member 3 (ENPP3) positive at pre-screening. This sub-group does not have any prior therapy requirement.
* Dose expansion cohorts: Histologically confirmed diagnosis of metastatic RCC of either clear cell or papillary histology

  * Tumors with clear cell histology: subject must have progressed after at least one anti-VEGFR therapy
  * Tumors with papillary histology: includes unclassified histology with papillary features and must be ENPP3 positive at pre-screening. This sub-group does not have any prior therapy requirement.
* Measurable disease according to Response Criteria for Solid Tumors (RECIST Version 1.1)
* Eastern Cooperative Group (ECOG) performance status of 0-1
* Hematologic function, as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL (transfusions are allowed)
* Renal function, as follows:

  * creatinine ≤ 1.5 x upper limit of normal (ULN), or calculated glomerular filtration rate (GFR) > 50 mL/min if creatinine > 1.5x ULN
* Hepatic function, as follows:

  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5x ULN if known liver metastases
  * Total bilirubin ≤1.5 x ULN
* International normalized ratio (INR) < 1.3 (or ≤ 3.0 if on therapeutic anticoagulation)
* Women and men of childbearing potential must be advised and agree to practice effective methods of contraception during the course of the study and for 4 weeks after the last AGS-16C3F infusion administration

Exclusion Criteria:

* Current uncontrolled central nervous system (CNS) metastasis or malignant brain tumors
* Use of any investigational drug (including marketed drugs not approved for this indication) within 4 weeks prior to screening. No time limit applies to the use of marketed drugs approved for this indication provided that the subject has progressed on the treatment and all toxicities attributable to the drug have resolved or returned to baseline
* Known sensitivity to any of the ingredients of the investigational product AGS-16C3F
* History of thromboembolic events and bleeding disorders ≤3 months (e.g., (deep vein thrombosis) DVT or pulmonary embolism (PE))
* Active angina or Class III or IV Congestive Heart Failure (CHF) (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by outpatient medication.
* Major surgery within 4 weeks of study enrollment
* Women who are pregnant (confirmed by positive pregnancy test) or lactating
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen.
* Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) within 72 hours of screening.
* History of eye surgery within 6 months, presence of cataracts or other ocular disorders significantly affecting vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07-18 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 24 months

SECONDARY OUTCOMES:
Pharmacokinetic profile for total antibody (TAb), antibody drug conjugate (ADC), and monomethyl auristatin F (MMAF): Ceoi or Cmax, Ctrough, Tmax, AUCτ, t1/2, CL, and Vss | Days 1, 2, 3, 4, 8, 15, 22, 43, 64, 65, 66, 67, 71, 78, and 92
  Concentration at end of infusion (Ceoi) or maximum observed concentrations (Cmax), Trough concentration (Ctrough), time to maximum concentration (Tmax), partial area under the serum concentration-time curve (AUCτ), terminal or apparent half-life (t1/2), systemic clearance (CL), and volume of distribution at steady state (Vss)
Incidence of antidrug antibody formation to human native antibody (AGS-16C) and antibody drug conjugate (AGS-16C3F) | 24 months
Tumor response: objective response rate | 24 months
  Determined from the subjects' best response and will include complete response (CR) and partial response (PR)
Tumor response: disease control rate | 24 months
  Determined from the subjects' best response will include complete response (CR) partial response (PR), and stable disease (SD)
Tumor response: Changes in bone scans | Baseline, Week 13 and every 12 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Agensys, Inc.
Locations (9):
- United States (5):
  - Site US00005 University of Michigan Medical Center, Ann Arbor, Michigan
  - Site US00003 Karmanos Cancer Institute, Detroit, Michigan
  - Site US00004 Roswell Park Cancer Institute, Buffalo, New York
  - Site US00002 Memorial Sloan-Kettering Cancer Center, New York, New York
  - Site US00001 Seattle Cancer Care Alliance, Seattle, Washington
- Canada (4):
  - Site CA00006 Cross Cancer Institute, Edmonton, Alberta
  - Site CA00008 British Columbia Cancer Agency, Vancouver, British Columbia
  - Site CA00009 London Health Sciences Centre, London, Ontario
  - Site CA00007 Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;AGS-16C3F-12-2